CLINICAL TRIAL: NCT00324194
Title: A Phase I Study of MGCD0103 Given as a Twice Weekly Oral Dose in Patients With Leukemia or Myelodysplastic Syndromes
Brief Title: A Phase I Study of MGCD0103 Given Twice Weekly in Patients With Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Gregory Reid, Chief Medical Officer, MethylGene, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-004
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: Leukemia; Myelodysplastic Syndromes; Phase I
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MGCD0103 oral dose 2 times per week.
  Interventions: Drug: MGCD0103

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 oral dose given 2 times per week.

SUMMARY:
In this study, MGCD0103, a new anticancer drug under investigation, is given twice weekly to patients with leukemia or myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of one of the following:

  * relapsed or refractory AML or ALL that has failed to respond to standard therapy, has progressed despite standard therapy.
  * relapsed or refractory Myelodysplastic Syndromes including CMML (chronic myelomonocytic leukemia) or other myeloproliferative disorders provided there is an MDS component.
  * previously untreated AML or Myelodysplastic Syndromes in patients >60 years of age who refused or are not candidates for induction chemotherapy
  * Patients with relapsed or refractory CML that has failed to respond to imatinib therapy or standard therapy, has progressed despite standard therapy, or for which no standard therapy exists.
* ECOG performance status of 0, 1, or 2.
* Age ≥18 years.
* Laboratory requirements.
* Patients or their legal representative must be able to read, understand, and sign a written informed consent (approved by the IRB/EC) prior to study entry.

Exclusion Criteria:

* Patients with other active malignancy except basal cell carcinoma or cervical intraepithelial neoplasia (CIN / cervical in situ).
* Patients with suspicion of CNS involvement (tests are not required to rule out CNS involvement in the absence of signs or symptoms).
* Pregnant or lactating women. Women of child-bearing potential must have a negative serum pregnancy test documented within 7 days prior to registration on study.
* Patients and their partners, if either are of childbearing potential, not using adequate birth control measures throughout the course of the study. Both men and women enrolled on study must agree to use a medically acceptable effective form of contraception during the study and for 90 days following the last dose of study medication. An effective form of contraception is an oral contraceptive or a double barrier method, such as condom with diaphragm.
* Patients with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results.
* Patients who have been treated with any investigational drug within 30 days prior to study initiation (an investigational drug is one for which there is no approved indication), or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy.
* Known hypersensitivity to any of the components of MGCD0103.
* Known HIV or Hepatitis B or C (tests do not need to be performed to rule out any of these infections).
* Any psychiatric illness/social situations that would, in the judgment of the investigator, limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-02; Primary Completion 2008-03 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability. | 1 year (anticipated)

SECONDARY OUTCOMES:
Clinical response. | 1 year (anticipated)
Dose limiting toxicities | 1 year (anticipated)
Pharmacokinetics | 1 year (anticipated)
Pharmacodynamics (histone acetylation, biomarkers) | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (4):
- United States (3):
  - Lee Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Columbia University Medical Center, New York, New York
- Sir Mortimer Davis Jewish General Hospital, Montreal, Quebec, Canada